CLINICAL TRIAL: NCT02209272
Title: Local Anesthesia for Ultrasound Guided Hip Joint Injections: A Double-Blinded Randomized Controlled Trial of Bacteriostatic Saline Versus Buffered Lidocaine
Brief Title: Comparison of Bacteriostatic Saline to Buffered Lidocaine for Ultrasound Guided Hip Joint Injection Local Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jacob L. Sellon, M.D., Assistant Professor of Physical Medicine and Rehabilitation, Sports Medicine Center, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-002622
Record Dates: First submitted 2014-07-31; First posted 2014-08-05 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Hip Pain
MeSH Terms: interventions — Benzyl Alcohol; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bacteriostatic saline (Experimental): for ultrasound guided hip joint injection local anesthesia
  Interventions: Drug: bacteriostatic saline
- buffered lidocaine (Active Comparator): for ultrasound guided hip joint injection local anesthesia
  Interventions: Drug: buffered lidocaine

INTERVENTIONS:
Drug: bacteriostatic saline
  Other Names: 0.9% benzyl alcohol
  Arms: bacteriostatic saline
Drug: buffered lidocaine
  Other Names: 1% lidocaine combined (9:1) with sodium bicarbonate
  Arms: buffered lidocaine

SUMMARY:
The purpose of this study is to compare infiltration pain and anesthetic efficacy between lidocaine and Bacteriostatic saline (BS) for ultrasound (US) guided intraarticular hip injections.

DETAILED DESCRIPTION:
Local anesthesia is commonly used to reduce pain during joint injections, particularly for deep joints like the hip. Lidocaine is the most commonly used local anesthetic in most medical practices. It is well known that lidocaine infiltration itself is painful. Many strategies have been studied to minimize pain associated with lidocaine administration, including buffering, warming, and slowing infiltration rate. BS is an alternative local anesthetic that has been shown to be less painful when injected into subcutaneous tissues compared with lidocaine. However, BS use has not been widely implemented for local anesthesia, and it has not been studied in the context of joint injections.

ELIGIBILITY:
INCLUSION CRITERIA:

* age 18-75 years
* referred for US-guided intraarticular hip injections in the Mayo Clinic Sports Medicine Center, Physical Medicine & Rehabilitation Clinic, or Musculoskeletal Clinic

EXCLUSION CRITERIA:

* chronic opioid use
* opioid use on day of procedure
* history of fibromyalgia or other diffuse chronic pain syndrome
* pain behavior during the clinical encounter as judged by the injectionist
* anesthetic administration time outside the designated 5-15 second time frame

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-08; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sellon, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Bacteriostatic Saline: In this arm patients received 2 injections:
  1. one injection of bacteriostatic saline (0.9% benzyl alcohol) in the skin, subcutaneous tissue and muscle overlying the hip joint using a 25 gauge needle
  2. a subsequent hip joint injection with corticosteroid and ropivacaine using a 22 gauge needle
  VAS-pain scores were collected immediately after each injection.
- Buffered Lidocaine: In this arm patients received 2 injections:
  1. one injection of buffered 1% lidocaine in the skin, subcutaneous tissue and muscle overlying the hip joint using a 25 gauge needle
  2. a subsequent hip joint injection with corticosteroid and ropivacaine using a 22 gauge needle
  VAS-pain scores were collected immediately after each injection.
Period: Overall Study
Arm/Group | Bacteriostatic Saline | Buffered Lidocaine
Started | 32 | 36
Completed | 32 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bacteriostatic Saline | Buffered Lidocaine | Total
Number analyzed (Participants) | 32 | 36 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (16) | 55.6 (16.1) | 54.9 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 23 | 40
  Male | 15 | 13 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 36 | 68

OUTCOME MEASURES:

1. Primary Outcome: VAS for Pain Score During Local Anesthesia Infiltration
Description: The Visual Analog Scale (VAS) for Pain is a validated tool used to measure pain. A 100mm horizontal line anchored by "no pain" (score of 0) and "pain as bad as it could be" (score of 100).
Time Frame: baseline to 5-10 minutes later -- immediately after local anesthetic injection administration
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Bacteriostatic Saline: for ultrasound guided hip joint injection local anesthesia
  bacteriostatic saline
- Buffered Lidocaine: for ultrasound guided hip joint injection local anesthesia
  buffered lidocaine
Arm/Group | Bacteriostatic Saline | Buffered Lidocaine
Number analyzed (Participants) | 32 | 36
score on a scale | 13.2 (15) | 14 (13.5)
Statistical Analysis 1: Comparison: Bacteriostatic Saline vs Buffered Lidocaine; Test type: Superiority; p = 0.82, t-test, 2 sided

2. Secondary Outcome: VAS for Pain Score During Subsequent Hip Joint Injection (Local Anesthetic Efficacy)
Description: as for outcome 1
Time Frame: baseline to 5-10 minutes later -- immediately after hip joint injection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bacteriostatic Saline | Buffered Lidocaine
Number analyzed (Participants) | 32 | 36
score on a scale | 20.7 (18.4) | 15.6 (13.9)
Statistical Analysis 1: Comparison: Bacteriostatic Saline vs Buffered Lidocaine; Test type: Superiority; p = 0.21, t-test, 2 sided

3. Secondary Outcome: Anesthetic Infiltration Duration
Description: Anesthetic infiltration duration will be measured using a timer on the ultrasound machine, with goal administration between 20-40 seconds.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Bacteriostatic Saline | Buffered Lidocaine
Number analyzed (Participants) | 32 | 36
seconds | 33.3 (4.5) | 32.7 (5)
Statistical Analysis 1: Comparison: Bacteriostatic Saline vs Buffered Lidocaine; Test type: Superiority; p = 0.57, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The study treatment follow-up period is defined as two weeks post-procedure.
Arm/Group | Bacteriostatic Saline | Buffered Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/36
Other Adverse Events (participants affected / at risk) | 0/32 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT02209272/Prot_SAP_000.pdf